CLINICAL TRIAL: NCT00724438
Title: Pharmacokinetics of Implanon in Obese Women
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: 15956A
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Contraception; Obesity
Keywords: Contraception; Implanon; Obesity; Blood spots; Implant; Pharmacokinetics
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Obese women: women with a body mass index (BMI) >30
- 2: Normal weight women: women with a BMI <25

SUMMARY:
Prior studies examining the pharmacokinetics, safety, and efficacy of the new etonogestrel-containing single rod implantable contraceptive device, Implanon, did not include women who exceeded 130% of ideal body weight. Yet, as these women comprise a significant portion of the U.S. population, studies of Implanon in obese women are essential. The proposed study represents an important first step in addressing the lack of data on Implanon in obese women. We aim to examine the pharmacokinetics of Implanon in obese women during the first 6 months of use and to provide data on the acceptability, side effect profile, and ease of insertion, palpation, and removal in these women. We also aim to collect samples for future validation studies of the use of the blood spot (finger-stick blood sample on filter paper) as a method of determining plasma etonogestrel.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal with a uterus and at least one ovary
* willing and able to sign the informed consent
* willing to comply with the study protocol and visit schedule
* have a body mass index of less than 25, or greater than or equal to 30
* weight stable

Exclusion Criteria:

* known or suspected pregnancy
* delivery (vaginal or cesarean) within 4 months of device insertion
* abortion (first or second trimester) within 4 months of device insertion
* contraindications to Implanon use
* hemophilia
* undiagnosed abnormal genital bleeding
* hypersensitivity or allergy to any components of Implanon
* personal or family history of thrombosis or thromboembolic disorders
* hepatic tumors or active liver disease
* known or suspected carcinoma of the breast or history of breast cancer
* more that one cardiovascular risk factor such as hypertension or diabetes
* known history of PCOS, diabetes, or glucose abnormality
* present use or use within 2 months of device insertion of a CYP3A4 inducer
* breastfeeding women
* use of an investigational drug within 2 months of device insertion
* use of injectable contraception within 6 months of device insertion
* planning a pregnancy in the next 12 months
* known HIV infection
* smoking over the age of 35

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited from resident and faculty practices at the University of Chicago outpatient facilities and from the University of Chicago clinical trails database of past study participants.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2008-07; Primary Completion 2009-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To describe the pharmacokinetic profile of Implanon (etonogestrel) among obese women. | 6 months

SECONDARY OUTCOMES:
To describe ease of insertion and palpation of Implanon among obese women | 6 months
To describe bleeding patterns among obese users of Implanon | 6 months
To describe the acceptability of Implanon among obese women | 6 months
To describe the discontinuation rates, reason for discontinuation, and ease of removal in obese women who discontinue the device before or at the end of the 6 month study period | 6 months
To determine whether etonogestrel levels can be obtained from finger-stick blood spots | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Gilliam, MD, MPH, Principal Investigator — University of Chicago; Sara J Mornar, DO, Study Director — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States